CLINICAL TRIAL: NCT00919074
Title: Comparison of Double Wire Technique With Pancreatic Duct Stent Placement for Difficult Bile Duct Cannulation: a Randomized Clinical Trial
Brief Title: Comparison of Double Wire Technique With Pancreatic Duct Stent Placement for Difficult Bile Duct Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Northwestern University (Other); University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 08-0831
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography (ERCP); Bile Duct Cannulation
Keywords: Patients undergoing endoscopic retrograde cholangiopancreatography for the first time; Particular focus on patients who meet predefined criteria for a difficult bile duct cannulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pancreatic duct stent (Active Comparator): Placement of a pancreatic duct stent to facilitate bile duct cannulation
  Interventions: Procedure: Pancreatic duct stent
- Pancreatic wire (Active Comparator): Placement of a guidewire into the pancreatic duct to facilitate bile duct cannulation.
  Interventions: Procedure: Pancreatic wire placement

INTERVENTIONS:
Procedure: Pancreatic duct stent — Placement of a pancreatic duct stent to facilitate bile duct cannulation
  Arms: Pancreatic duct stent
Procedure: Pancreatic wire placement — Placement of a pancreatic wire to facilitate bile duct cannulation
  Arms: Pancreatic wire

SUMMARY:
This research project will compare the use of the double wire technique with the placement of a pancreatic duct (PD) stent to achieve deep biliary cannulation without the use of a precut papillotomy. Currently, the data supporting either of these approaches is limited to the referenced case series. More data on the success and complication rates of these techniques are needed. The investigators believe either of these approaches would be preferred by less experienced endoscopists to precut papillotomy. Consequently, it is important to differentiate these techniques and identify which patients may benefit from one or both.

ELIGIBILITY:
Inclusion Criteria:

* First time ERCP

Exclusion Criteria:

* Successful bile duct cannulation within six minutes
* Planned pancreatic duct therapy
* Planned pancreatobiliary manometry
* Prior successful ERCP

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2008-09; Primary Completion 2011-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Cannulation success rate | Cannulation is assessed during the index procedure; procedure-related complications are assessed within one week of the procedure

SECONDARY OUTCOMES:
Complication rate | One week

CONTACTS AND LOCATIONS:
Overall Officials: Riad R Azar, MD, Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - Washington University in St. Louis, St Louis, Missouri
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma

REFERENCES:
- [Result] Cote GA, Mullady DK, Jonnalagadda SS, Keswani RN, Wani SB, Hovis CE, Ammar T, Al-Lehibi A, Edmundowicz SA, Komanduri S, Azar RR. Use of a pancreatic duct stent or guidewire facilitates bile duct access with low rates of precut sphincterotomy: a randomized clinical trial. Dig Dis Sci. 2012 Dec;57(12):3271-8. doi: 10.1007/s10620-012-2269-2. Epub 2012 Jun 26. PMID 22732831